CLINICAL TRIAL: NCT01143350
Title: Non Pharmacological Treatment in Alzheimer's Disease and Associated Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: CAILLON Cynthia, DRCI du CHU de Nice
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 09-PP-09
Record Dates: First submitted 2010-02-25; First posted 2010-06-14 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2010-03

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- EHPAD Training and Stimulation (Experimental): EHPAD of the group of Training / Stimulation will benefit:
  * after a training in behaviours to be held or in methods of stimulation aiming at the reduction of disturbances of behaviour at type of apathy. This information will be transmitted in l 'ensemble of l 'équipe of l 'EHPAD by a training officer.
  * of a structuring of the activities of animation offered to the inhabitants, This information will be regrouped in chips worked out like TNM - EHPAD.
  Interventions: Other: Bras A (EHPAD Training and stimulation)
- 2- EHPAD control (Placebo Comparator): EHPAD of the reference group, will have their habitual functioning
  Interventions: Other: EHPAD Control

INTERVENTIONS:
Other: Bras A (EHPAD Training and stimulation) — EHPAD of the group of Training / Stimulation will benefit:
  * after a training in behaviours to be held or in methods of stimulation aiming at the reduction of disturbances of behaviour at type of apathy. This information will be transmitted in l 'ensemble of l 'équipe of l 'EHPAD by a training officer.
  * of a structuring of the activities of animation offered to the inhabitants, This information will be regrouped in chips worked out like TNM - EHPAD.
  Arms: EHPAD Training and Stimulation
Other: EHPAD Control — EHPAD of the reference group, will have their habitual functioning
  Arms: 2- EHPAD control

SUMMARY:
The STIM-EHPAD study (for stimulation in nursing home) aims to evaluate the short and medium term effectiveness of staff education as a non-pharmacological intervention to manage apathy in older people with a diagnosis of dementia.

* Primary efficacy criteria: Apathy Inventory clinician score changes
* Secondary efficacy criteria: Apathy Inventory patient and caregiver version changes, Observation scale changes, frequency and severity of the other BPSD using the NPI, qualitative analysis of the nursing home staff behavioural changes

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 65 years
* A diagnosis of dementia according to the ICD 10 criteria
* MMSE score ≤ 24
* Presenting the diagnostic criteria of apathy (cf page ??)
* An Apathy Inventory clinician total score >3 (with at least a score higher than 1 at one of the 3 dimensions; lack of initiative, lack of interest, emotional blunting)

Exclusion Criteria:

* Patients more than 65 years
* MMSE score > 24

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Identification of yet unknown enzymes involved in the processing of Ab, especially on those responsible for the exoproteasic truncation of Ab at its N-terminus. | 1 year
  Identification of yet unknown enzymes involved in the processing of Ab, especially on those responsible for the exoproteasic truncation of Ab at its N-terminus.

SECONDARY OUTCOMES:
Secondary efficacy criteria: Apathy Inventory patient and caregiver version changes, Observation scale changes, frequency and severity of the other BPSD using the NPI, qualitative analysis of the nursing home staff behavioural changes | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Ph ROBERT, PhD, Principal Investigator — CHU de Nice - CM2R - Hôpital de Cimiez - 4 avenue reine victoria - 06 003 Nice cedex 1
Locations (1):
- Robert, Nice, Alpes-Maritimes, France